CLINICAL TRIAL: NCT03661255
Title: Promoting Community Conversations About Research to End Native Youth Suicide in Rural Alaska
Acronym: PC CARES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Nebraska Lincoln (Other); Norton Sound Health Corporation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Wexler, Professor of Social Work, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00161969; 1R01MH112458-01A1 (NIH)
Record Dates: First submitted 2018-07-12; First posted 2018-09-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Suicide
Keywords: Suicide Prevention; Alaska Native; Community Intervention
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: The study will have a stepped wedge design with 3 cohorts (in successive years) of 3 villages each. In each village, we will collect baseline data and follow-up data on knowledge, attitudes, and behavior related to suicide prevention from participants and non-participants. Participants will also provide data on these topics after each learning circle they attend. Intervention participants will be self-selecting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC CARES Intervention (Experimental): Experimental: PC CARES Intervention Participants will attend 1-7 sessions of the PC CARES curriculum, either virtually or in-person. Investigators will collect data from this group at baseline, after each session they attend, and at follow-up.
  Interventions: Behavioral: PC CARES
- No intervention (No Intervention): This group will not attend the PC CARES sessions. Investigators will collect data from this group at baseline and follow-up

INTERVENTIONS:
Behavioral: PC CARES — PC CARES trains local residents to deliver the PC CARES curriculum in their own community. These facilitators will attend a 40 hour training, and then will deliver the 4 session PC CARES curriculum in their home village. To aid local facilitators, each session follows the same structure after a beginning ritual:(1) agreements/safe talk, (2)'small wins', (3)'what do we know?' (facilitator shares current research on suicide prevention or wellness) (4)'what do we think?' (participants have an opportunity to discuss their thoughts on the research presented), and (5)'what we want to do?' (participants identify what steps they can take in their village to make positive change).The content of learning circles (LCs) includes community-level conditions, evidence-based approaches, risk and protective factors that can prevent suicide and promote well-being.Each LC includes both primary and secondary prevention strategies.Teaching tools include charts, short films, and case studies.
  Arms: PC CARES Intervention

SUMMARY:
This intervention study measures the outcomes of the PC CARES (Promoting Community Conversations about Research to End Suicide) project implemented in remote rural Alaskan villages. Researchers worked with local service providers and other partners to recruit facilitators who were trained to implement the 5-session PC CARES curriculum. The study will compare pre-post data from intervention participants to non-participants, and will analyze social networks related to suicide prevention behavior in each village.

DETAILED DESCRIPTION:
This intervention study will measure the outcomes of the PC CARES (Promoting Community Conversations about Research to End Suicide) curriculum implemented in 9 rural Alaskan villages and remotely during COVID pandemic years (2020-2022). It will compare pre-post data from intervention participants to non-participants, and will analyze social networks related to suicide prevention behavior in each village. Researchers worked with local service providers and other partners to recruit participants who have access to the internet for virtual sessions. Pilot research by the investigators produced a roster of social ecological roles within the village (hereafter: 'network positions') that are relevant to suicide prevention. These network positions include organizational affiliations: individuals interacting with young people as a function of their position in schools, health care facilities, mental health services, social services, religious institutions, tribal governments, city governments (including law enforcement). The roster also includes family roles: Elder; parent; a sibling or cousin who is close; other adult family member who is also a mentor: or friend. Mainly school-based personnel and clinic-based staff were recruited to attend the 7 virtual PC CARES sessions.

Baseline data collection:

For pre-intervention data collection, investigators recruited widely in each village, focusing on those who occupy organizationally-affiliated network positions, and youth ages 15-24. Data collection will involve a survey in which they will be asked about demographics, Knowledge about reducing suicide, Skills in making positive community changes, Attitudes toward suicide prevention, and Behavior related to suicide prevention. Questions about Behavior included follow up questions asking with whom they've done the behavior (which of the listed network positions) and 'How Often?'

The study's original Interrupted Time Series design had 3 cohorts, with the opportunity for all villages in the Bering Strait region of Alaska to participate. However, the COVID-19 pandemic led to modifications to: 1) the intervention delivery method, 2) audience, and 3) content. After the first cohort of in-person learning circles was halted to follow health authority guidelines, PC CARES pivoted to 1) online, remote synchronous delivery (live Zoom sessions) with 2) school and clinic staff in any of the Bering Strait region and Northwest Arctic region communities (27 villages total), with 3) additional sessions regarding school-specific suicide prevention strategies. Schools are some of the best-resourced institutions in the villages, with existing infrastructure like wireless Internet and spaces for community use, and school staff are well-positioned to make impacts on youth wellness.

During COVID, we offered online, all-staff 'one time' inservice trainings for Bering Strait School District and Northwest Arctic School District staff on what they can do (and the school as a whole can do) to prevent suicide among their students. Afterward, interested staff and community members were invited to participate in on-going virtual learning circles hosted by PC CARES curriculum trainers aimed at developing a suicide prevention and postvention plan for their school and/or district. School staff who were at least 18 years old, and who participated in any level of training will have the option to participate in 3 online surveys (emailed to them) to assess their changes in Attitudes, Skills, Behavior, Knowledge and Community of Practice related to suicide prevention: 1) before any trainings are offered, 2) soon after the inservice, and 3) at the end of the school year.

Participants in the Virtual PC CARES training filled out a registration form to indicate their interest in attending PC CARES. The registration form included a description of the research and consent form. If they gave their informed consent, participants were brought to the Virtual PC CARES Baseline Survey, which mirrors the Steps Toward Prevention Survey, with a few questions that pertain to the school context added. We also added some answer choices for school-specific network roles such as Teacher, Administrator, Coach, Administrative Assistant/Front Desk, Classroom Aide, Other school staff (including janitor/cafeteria worker), Student, Parent of student. Participants in the virtual sessions were asked for their consent to use the notes from PC CARES sessions as part of the research. Students who did not consent were excluded from note-taking.

Also due to COVID-related restrictions, we began to send PC CARES Care packages to community members who 'opted in' to receive them. Care packages contained brief information about what research shows community members can do to prevent suicide and promote wellness in their community. They will also contain small gifts that community members can use in their wellness promotion/suicide prevention, such as "You Matter" cards that have affirming messages that they can share with others in their community. Over 2 years, PC CARES sent Care Packages to 493 recipients in 49 communities in Alaska, with a total number of 1319 packages sent. Each care package contained a survey with a self-addressed stamped envelope. Participants who sent the survey back to researchers or filled it out online were entered into a raffle to win a prize worth $50. After each care package, we also randomly selected 5 Care package recipients to be invited to participate in a brief interview to collect additional data about how they are using the Care package information and items and to help us make the Care packages more useful to them over time. Interview participants received a $20 gift card as an incentive to participate. According to recipient feedback, the Care Packages helped build connections and goodwill between PC CARES and participants during COVID-19 pandemic, and were welcomed and well-used by recipients.

As a supplement to the original grant and the virtual adaptation, we initiated an implementation-focused small study. In this additional project, a cohort of students in the Rural Human Services Certificate Program at University of Alaska-Fairbanks, Kuskokwim campus will fulfill their practicum requirement by facilitating PC CARES Learning Circles in their home communities in rural remote western Alaska. Students who consent to participate in the study will complete 3 surveys (Pre-Training, Post-Training, and 6-Month Follow Up). In addition, we asked for consent to take field notes during the facilitator training and during the monthly facilitator support calls. These field notes focus on what kinds of questions are raised by trainees, what challenges and success they have as facilitators, and other information related to the experience of being a facilitator.

Follow Up data collection:

For data collection approximately 1 month after the intervention concluded, investigators recruited all those who attended PC CARES and those who completed the baseline survey. This survey was identical to the Baseline Survey, and participants' responses were paired to their baseline data via anonymous IDs. By starting with those who attended PC CARES sessions, investigators hope to document diffusion effects-to learn how PC CARES impacts those who attend the learning circles, people close to them and others in the community.

Our expected recruitment numbers evolved as the ramifications of the COVID pandemic hit and our strategy had to change. Pre-pandemic, we were able to recruit 496 participants who completed a Baseline Steps toward Prevention Survey, however, we shifted our research strategy to hold virtual learning circles based in the schools in 2 remote Alaskan regions. With this revised scope, we aimed to recruit 700 and in actuality, we recruited 774.

Also due to COVID, we instated the PC CARES at Home Care Package program and we had 117 participants.

In our efforts to research further the experiences of PC CARES facilitators, we planned to recruit 20 students from the UAF-Bethel Rural Human Services program, and 24 of them have enrolled.

This study maximizes rigor through a multiple baseline, multi-method approach, and carefully tracks the process indicators, moderating variables, and mechanisms leading to our hypothesized proximal, intermediate and ultimate outcomes of youth support to reduce suicidal behavior. Most community-based suicide studies measure only changes in participants' knowledge, attitudes and intentions to act. This study goes further by documenting changes in participants' prevention behavior over time, and assessing its impact on protective interactions within the community.

Integrating key lessons from the pilot research, investigators use multilevel growth modeling to track the factors likely to affect these outcomes, namely participation at community (cross- sector) and individual (dosage) levels, and the formal/institutional or informal/community social role of participants. Using innovative social network methods, investigators also investigate the intervention's impact on prevention-oriented interactions, help- giving and seeking, and health promoting exchanges within the community.

By documenting the level and type of preventive and supportive interactions taking place among people in various roles (including youth) within the village before and after PC CARES, investigators can assess the effectiveness of the intervention at initiating community-level change among PC CARES participants and those who did not participate: allowing investigators to measure diffusion effects. This data informs investigators of the scalability of the approach. This analysis considers the moderating effects of key variables such as the degree of closeness between youth and PC CARES participants, level of collaboration between formal-informal supporters, interactions across age groups, and level of participation. Building on the infrastructure of schools and tribal health clinics in each rural and remote community and leveraging our prior work, our scalable model translates scientific prevention research onto practice, enabling people who are in the daily lives of Alaska Native youth to purposefully reduce suicide risk factors, and increase safety, help-seeking and support to prevent suicide and promote health.

ELIGIBILITY:
Inclusion Criteria:

* lives or works in village
* at least 15 years old

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1491 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Behaviors related to suicide prevention | 6 times over approximately 3 year period
  Behaviors (12 survey questions) related to suicide prevention will be measured at baseline, after each PC CARES session, and at follow up for participants (intervention group) and at baseline and followup only for non-participants (No intervention group).
Change in Knowledge related to suicide prevention | 6 times over approximately 3 year period
  Knowledge (7 survey questions) related to suicide prevention will be measured at baseline, after each PC CARES session, and at follow up for participants (intervention group) and at baseline and followup only for non-participants (No intervention group).
Change in Attitudes related to suicide prevention | 6 times over approximately 3 year period
  Attitudes (20 survey questions) related to suicide prevention will be measured at baseline, after each PC CARES session, and at follow up for participants (intervention group) and at baseline and followup only for non-participants (No intervention group).

SECONDARY OUTCOMES:
Community level impact of PC CARES (type of interactions) | Pre and post intervention (2 times over approximately 3 year period)
  Investigators will document the community level impact of PC CARES by tracking the type of interactions aimed at preventing youth suicide and promoting wellness in participating villages
Community level impact of PC CARES (number of interactions) | Pre and post intervention (2 times over approximately 3 year period)
  Investigators will document the community level impact of PC CARES by tracking the number of interactions aimed at preventing youth suicide and promoting wellness in participating villages
Community level impact of PC CARES through social network analysis by describing changes in the supportive social networks of young people before and after the intervention. | Pre and post intervention (2 times over approximately 3 year period)
  Document the Community level impact of PC CARES by describing changes in the supportive social networks of young people before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Wexler, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Final data will be shared through peer-reviewed publications and presentations, community presentations and tribal reports. Raw data will be considered for sharing under the following rules. Raw datasets released for sharing will not contain identifiers. Data and associated documentation will be made available to users only under a signed and properly executed data-sharing agreement that provides specific criteria under which the data will be used, including but not limited to: (1) a commitment to secure the data using appropriate computer technology, (2) a commitment to using the data for research purposes that are in accordance with collaborating tribes' priorities, (3) that the data is not used to identify individual participants and conforms to all privacy protections indicated in the participants' informed consent, and (4) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Wexler L, Trout L, Rataj S, Kirk T, Moto R, McEachern D. Promoting Community Conversations About Research to End Suicide: learning and behavioural outcomes of a training-of-trainers model to facilitate grassroots community health education to address Indigenous youth suicide prevention. Int J Circumpolar Health. 2017;76(1):1345277. doi: 10.1080/22423982.2017.1345277. PMID 28762305
- [Background] Wexler L, McEachern D, DiFulvio G, Smith C, Graham LF, Dombrowski K. Creating a Community of Practice to Prevent Suicide Through Multiple Channels: Describing the Theoretical Foundations and Structured Learning of PC CARES. Int Q Community Health Educ. 2016;36(2):115-22. doi: 10.1177/0272684X16630886. Epub 2016 Feb 15. PMID 26880738
- [Background] Lee HW, Gauthier GR, Ivanich JD, Wexler L, Khan B, & Dombrowski K. A method for assessing the success and failure of community-level interventions in the presence of network diffusion, social reinforcement, and related social effects. ArXiv180108612 Phys. January 2018. http://arxiv.org/abs/1801.08612. Accessed February 8, 2018.
- [Background] Palinkas LA, Holloway IW, Rice E, Brown CH, Valente TW, Chamberlain P. Influence network linkages across implementation strategy conditions in a randomized controlled trial of two strategies for scaling up evidence-based practices in public youth-serving systems. Implement Sci. 2013 Nov 14;8:133. doi: 10.1186/1748-5908-8-133. PMID 24229373
- [Background] Gest SD, Osgood DW, Feinberg ME, Bierman KL, Moody J. Strengthening prevention program theories and evaluations: contributions from social network analysis. Prev Sci. 2011 Dec;12(4):349-60. doi: 10.1007/s11121-011-0229-2. PMID 21728069
- [Background] Tseng V. The uses of research in policy and practice. Sharing Child and Youth Development Knowledge 26(2):1-16, 2012.
- [Background] Rogers EM. Diffusion of Innovations. NY, NY Simon and Schuster, 2010.
- [Background] Dombrowski K, Khan B, Moses J, Channell E, & Dombrowski N. Network sampling of social divisions in a rural Inuit community. Identities 21(2):134-151, 2014.
- [Background] Wexler LM. Inupiat youth suicide and culture loss: Changing community conversations for prevention. Soc Sci Med. 2006 Dec;63(11):2938-48. doi: 10.1016/j.socscimed.2006.07.022. Epub 2006 Sep 6. PMID 16952416
- [Background] Wexler L, Goodwin B. Youth and adult community member beliefs about Inupiat youth suicide and its prevention. Int J Circumpolar Health. 2006 Dec;65(5):448-58. doi: 10.3402/ijch.v65i5.18146. PMID 17319089
- [Background] Hill R, Perkins R, Wexler L. An analysis of hospital visits during the 12 months preceding suicide death in Northern Alaska. Alaska Med. 2007 Jan-Mar;49(1):16-21. PMID 17479732
- [Background] Wexler L, Hill R, Bertone-Johnson E, Fenaughty A. Correlates of Alaska Native fatal and nonfatal suicidal behaviors 1990-2001. Suicide Life Threat Behav. 2008 Jun;38(3):311-20. doi: 10.1521/suli.2008.38.3.311. PMID 18611129
- [Background] Wexler L. Identifying colonial discourses in Inupiat young people's narratives as a way to understand the no future of Inupiat youth suicide. Am Indian Alsk Native Ment Health Res. 2009;16(1):1-24. doi: 10.5820/aian.1601.2009.1. PMID 19340763
- [Background] Wexler L. Behavioral health services "Don't work for us": cultural incongruities in human service systems for Alaska Native communities. Am J Community Psychol. 2011 Mar;47(1-2):157-69. doi: 10.1007/s10464-010-9380-3. PMID 21052820
- [Background] Ulturgasheva O, Wexler L, Kral M, Allen J, Mohatt GV, Nystad K; CIPA Team. Navigating International, Interdisciplinary, and Indigenous Collaborative Inquiry: Phase 1 in the Circumpolar Indigenous Pathways to Adulthood Project. J Community Engagem Scholarsh. 2011 Jun 19;4(1):50-59. PMID 22866196
- [Background] Wexler L, Silveira ML, Bertone-Johnson E. Factors associated with Alaska Native fatal and nonfatal suicidal behaviors 2001-2009: trends and implications for prevention. Arch Suicide Res. 2012;16(4):273-86. doi: 10.1080/13811118.2013.722051. PMID 23137218
- [Background] Wexler L, Gubrium A, Griffin M, DiFulvio G. Promoting positive youth development and highlighting reasons for living in Northwest Alaska through digital storytelling. Health Promot Pract. 2013 Jul;14(4):617-23. doi: 10.1177/1524839912462390. Epub 2012 Oct 24. PMID 23099660
- [Background] Wexler L, Jernigan K, Mazzotti J, Baldwin E, Griffin M, Joule L, Garoutte J Jr; CIPA Team. Lived challenges and getting through them: Alaska Native youth narratives as a way to understand resilience. Health Promot Pract. 2014 Jan;15(1):10-7. doi: 10.1177/1524839913475801. Epub 2013 Feb 21. PMID 23431127
- [Background] Wexler L. Looking across three generations of Alaska Natives to explore how culture fosters indigenous resilience. Transcult Psychiatry. 2014 Feb;51(1):73-92. doi: 10.1177/1363461513497417. Epub 2013 Sep 6. PMID 24014514
- [Background] Wexler L, Joule L, Garoutte J, Mazziotti J, Hopper K. "Being responsible, respectful, trying to keep the tradition alive:" cultural resilience and growing up in an Alaska Native community. Transcult Psychiatry. 2014 Oct;51(5):693-712. doi: 10.1177/1363461513495085. Epub 2013 Sep 6. PMID 24014513
- [Background] Allen J, Hopper K, Wexler L, Kral M, Rasmus S, Nystad K. Mapping resilience pathways of Indigenous youth in five circumpolar communities. Transcult Psychiatry. 2014 Oct;51(5):601-31. doi: 10.1177/1363461513497232. Epub 2013 Aug 21. PMID 23965730
- [Background] Ulturgasheva O, Rasmus S, Wexler L, Nystad K, Kral M. Arctic indigenous youth resilience and vulnerability: comparative analysis of adolescent experiences across five circumpolar communities. Transcult Psychiatry. 2014 Oct;51(5):735-56. doi: 10.1177/1363461514547120. PMID 25217145
- [Background] Wexler L, Chandler M, Gone JP, Cwik M, Kirmayer LJ, LaFromboise T, Brockie T, O'Keefe V, Walkup J, Allen J. Advancing suicide prevention research with rural American Indian and Alaska Native populations. Am J Public Health. 2015 May;105(5):891-9. doi: 10.2105/AJPH.2014.302517. Epub 2015 Mar 19. PMID 25790403
- [Background] Silveira ML, Wexler L, Chamberlain J, Money K, Spencer RM, Reich NG, Bertone-Johnson ER. Seasonality of suicide behavior in Northwest Alaska: 1990-2009. Public Health. 2016 Aug;137:35-43. doi: 10.1016/j.puhe.2016.02.010. Epub 2016 Mar 24. PMID 27021788
- [Background] Curran T, Wexler L. School-Based Positive Youth Development: A Systematic Review of the Literature. J Sch Health. 2017 Jan;87(1):71-80. doi: 10.1111/josh.12467. PMID 27917486
- [Background] Hagan K, Hill R, & Wexler L. The prevention of suicide within the Health Care setting and in Alaska. Primary Care:Indian Health Service, 32(7):198-201, 2007.
- [Background] Wexler L, & Graves K. The importance of culturally-responsive training for building a behavioral health workforce in Alaska Native villages: A case study from Northwest Alaska. Special SAMHSA issue of the Journal of Rural Mental Health 32(3): 22-33, 2008.
- [Background] Wexler L. The importance of identity, culture and history in the study of indigenous youth wellness. The Journal of the History of Childhood and Youth 2(2):267-278, 2009.
- [Background] Wexler L. Intergenerational exchange as data collection: introducing a community-based participatory approach to connect youth, adults and elders in a tribal community. International Journal of Qualitative Methods 10(3): 248-264, 2011.
- [Background] Wexler LM, Gone JP. Culturally responsive suicide prevention in indigenous communities: unexamined assumptions and new possibilities. Am J Public Health. 2012 May;102(5):800-6. doi: 10.2105/AJPH.2011.300432. Epub 2012 Mar 15. PMID 22420786
- [Background] Wexler L, Eglinton K, & Gubrium A. Using digital stories to understand the lives of Alaska Native young people. Youth & Society 46(4): 478-504, 2014.
- [Background] Wexler L, White J, Trainor B. Why an alternative to suicide prevention gatekeeper training is needed for rural Indigenous communities: presenting an empowering community storytelling approach. Crit Public Health. 2015;25(2):205-217. doi: 10.1080/09581596.2014.904039. Epub 2014 Apr 7. PMID 36779086
- [Background] Wexler L & Gone JP. Exploring alternatives for Indigenous suicide prevention: Responding to cultural understandings and practices. In Jennifer White, Ian Marsh, Michael Kral & Jonathan Morris (Eds), [Suicide and] Suicide Prevention: Critical Perspectives, Cambridge University Press, 2015.
- [Background] Wexler L, Dam HT, Silvius K, Mazziotti J, &Bamikole I. Protective factors of Native youth: findings from a self-report survey in rural Alaska. Journal of Youth Studies 19(3): 358-373, 2016.
- [Background] Wexler L, Poudel-Tandukar K, Rataj S, Trout L, Poudel KC, Woods M, Chachamovich E. Preliminary Evaluation of a School-Based Youth Leadership and Prevention Program in Rural Alaska Native Communities. School Ment Health. 2017 Jun;9(2):172-183. doi: 10.1007/s12310-016-9203-2. Epub 2016 Nov 19. PMID 35572790
- [Background] White LA, Wexler L, Weaver A, Moto R, Kirk T, Rataj S, Trout L, McEachern D. Implementation beyond the clinic: Community-driven utilization of research evidence from PC CARES, a suicide prevention program. Am J Community Psychol. 2022 Dec;70(3-4):365-378. doi: 10.1002/ajcp.12609. Epub 2022 Jun 28. PMID 35762450
- [Background] Wells CC, White L, Schmidt T, Rataj S, McEachern D, Wisnieski D, Garnie J, Kirk T, Moto R, Wexler L. Adapting PC CARES to Continue Suicide Prevention in Rural Alaska During the COVID-19 Pandemic: Narrative Overview of an In-Person Community-Based Suicide Prevention Program Moving Online. Am Indian Alsk Native Ment Health Res. 2022;29(2):126-154. doi: 10.5820/aian.2902.2022.126. PMID 35881985
- [Background] Markowski KL, White L, Harcey SR, Schmidt T, McEachern D, Habecker P, Wexler L. What Kinds of Support are Alaska Native Youth and Young Adults Reporting? An Examination of Types, Quantities, Sources, and Frequencies of Support. Health Promot Pract. 2023 Sep;24(5):863-872. doi: 10.1177/15248399221115065. Epub 2022 Sep 1. PMID 36047453
- [Background] Wexler L, Schmidt T, White L, Wells CC, Rataj S, Moto R, Kirk T, McEachern D. Collaboratively adapting culturally-respectful, locally-relevant suicide prevention for newly participating Alaska Native communities. Journal for Social Action in Counseling and Psychology. 2022; 14(1): 124-151. https://doi.org/10.33043/JSACP.14.1.124-151
- See also: Site describing the PC CARES philosophy, curriculum, team, and how people can get involved — http://www.pc-cares.org/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03661255/Prot_SAP_ICF_002.pdf